CLINICAL TRIAL: NCT06091111
Title: A Clinical Trial to Evaluate Leakage Performance in a Hybrid Absorbing Incontinence Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Collaborators: Lincolnshire Community Health Services NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HEAT
Record Dates: First submitted 2023-10-12; First posted 2023-10-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Single group cross over. Study subjects are randomized to sequence of device use. To either start with reference of study device.
Masking Description: As the study device is obviously different to the currently used device, and all subjects will use the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental): Subjects is randomized to start with either a period of reference product use followed by a cross over to using the study device or the opposite sequence, starting with the study device and then cross over to using the reference device.
  Interventions: Device: THD, THN

INTERVENTIONS:
Device: THD, THN — New hybrid absorbing incontinence product for day (THD) and night (THN) use. These are variants of the same product. The intervention product is a novel design that contains reusable elements allowing for a more sustainable product.

SUMMARY:
The study is prospective, sequential, single group, and interventional but not invasive. The primary objective is to evaluate the leakage performance of the investigational medical devices (absorbing hygiene products, AHPs) compared to reference AHPs currently being used by the subjects. The study is cross-over and subjects will act as their own control, using their regular device during a 10-day period and comparing this to use of investigational device for 10 days with an initial 3-5 day transition period. In total the subjects participate in the study for about 30 days. The sequence of device use is randomized. The target population are subjects who are suffering from urinary incontinence and are current users of AHPs to manage the incontinence. Subjects are care dependent and being cared for in a care home. The study is conducted at multiple care homes in the United Kingdom. The investigational device is a new type of AHP developed to be more sustainable with a disposable insert placed into a reusable pant. The leakage performance will be tracked by collecting used AHPs and assess the occurrence of leakages and urine content. The number of leakages during the intervention period will be compared to that of the reference period. As secondary outcomes safety, changes in skin condition and caregiver and subject product satisfaction is assessed. In total 42 subjects are planned for the study.

DETAILED DESCRIPTION:
This is a pre-market feasibility clinical investigation designed to evaluate the clinical performance and safety of the investigational product in its intended target population.

The clinical investigation is designed according to the ISO 14155:2020 to be prospective, interventional but non-invasive, at multiple care homes and randomised.

There is one group using two different reference products (TENA Comfort or TENA Slip) Cross-over with randomised sequential product use. Use of reference product (TENA comfort or TENA Slip) and investigational product (THD and THN) use.

Residents uses regular (reference) product for 10 days and then switch to the investigational product and use it for 10 days. There will be a 3-5-day transition period when the investigational product is introduced and then follows the 10-day evaluation period.

The investigational and the reference products for this study are absorbing hygiene products (class I medical devices) used as urine incontinence aids. Investigational devices (products) are new specifications THD and THN. THD and THN are hybrid products, consisting of a single use insert and a reusable pant, developed to be more sustainable than the current products in the market. Reference products are current all-in-one and/or two-piece product on the market TENA Slip/Comfort with super, plus and maxi absorption level and sizes M and L.

Primary objective: To evaluate the leakage performance of the investigational products compared to reference products.

Secondary objective(s):

To evaluate safety through analysing product-related adverse events reported during the investigation.

To evaluate any changes in skin condition of the resident during the course of the investigation.

To evaluate caregiver and subject, satisfaction, perception of and experience in using the products related to comfort, softness, dryness, skin health and ease of product washing.

In the study, the products are used by individuals, residents, suffering from incontinence who are cared for in a care home, by one or more professional caregivers.

Multiple care homes within Lincolnshire in the United Kingdom. Lincolnshire Community Health Services National Health Services Trust acts as site and coordinates the care homes. Care homes will be randomised to either start with reference product or investigational product.

A total of 42 subjects is to be included.

For the residents there will be 5 visits:

Visit 1 Screening and recruitment. Visit 2 Period 1 start (Day 0). Visit 3 Transition period start (Day 10+3). Visit 4 Start of period 2 (3-5 days after visit 3). Visit 5 Study completion (Day 10+3 after visit 4).

Between visit 2 and 5 there will be a daily collection by the study team of labelled bags containing used products. These products will then be weighed, labels retrieved, and photos taken.

A descriptive analysis will be carried out for all variables and endpoints. For the analysis each tested product is classified according to presence of leakage (Yes/No). The proportion of products that do not leak is designated the success rate (SR). A non-inferiority one-sided paired t-test will be performed to analyse the primary endpoint.

For the safety endpoint, data on incidence and severity of adverse events related to products will be summarized.

The error rate is set to 2.5% for the primary endpoint and 5% for secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Have urinary incontinence managed with size M or L (96 -116 cm hip range) TENA Slip and/or TENA Comfort with absorption level plus, super or maxi.
* Be willing and able to provide informed consent and to participate in the clinical investigation.
* Be a permanent (intended length of stay longer than 3 months) resident of the care home.
* Have a stable dose regime if the incontinence is managed by pharmaceuticals.
* Be over 18 years of age.
* Not be of child-bearing potential.

Exclusion Criteria:

* Being cared for at home or outside of professional care environment.
* Goes to the toilet to urinate regularly.
* Have severe incontinence product related skin problems, as judged by the investigator.
* Have any type of urinary catheter(s) resulting in improved/treated urinary incontinence.
* Suffering from fecal incontinence with a severity that makes participation in the clinical investigation inappropriate, as judged by investigator.
* Suffer from severe dementia that makes participation in the clinical investigation inappropriate, as judged by investigator.
* Having any other condition or recent surgery that may make participation in the clinical investigation inappropriate, as judged by investigator.
* Frequently removes the incontinence product by themselves.
* Have participated in an investigational study of a drug, biologic, or medical device within 30 days prior to entering the clinical investigation or planned during the clinical investigation.
* Having an alcohol or drug addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in absorbing product leakage rate | 20 days
  For each resident a success rate (SR, number of products that do not have a urine leakage outside of the product) is calculated and compared between the baseline (standard of care) and the intervention (study device).

SECONDARY OUTCOMES:
Safety data | 20 days
  Incidence of adverse events (AE), adverse product effects (ADE), serious adverse events (SAE), serious adverse device effects (SADE), and device deficiency (DD).
Skin health assessment scoring. | 20 days
  The skin health is followed via a scoring for incontinence associated dermatitis (IAD). The scoring between baseline and intervention are compared. The scoring is on 1-5 scale for grading the skin injury were 1 is no skin irritation and 5 severe skin irritation with infection. Also there is an overall skin problem scoring on a 1-5 scale were 1 is none and 5 is very severe.
Caregiver and resident scoring perception of the investigational product compared to the reference product. | 20 days
  Questionnaire with question regarding the perception and satisfaction of the investigational device regarding some specific aspects like comfort, ease of use and feeling on the skin. The scoring is made for each aspect based on a 1-5 Likert scale were 5 represents the highest value.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Weisman, Principal Investigator — Lincolnshire Community Health Services NHS
Locations (1):
- Lincolnshire Community Health Services NHS Trust, Lincoln, United Kingdom

IPD SHARING:
Plan to Share IPD: No